CLINICAL TRIAL: NCT01572792
Title: A Phase III, Long-term, Randomized, Double-blind, Extension Study of the Efficacy, Safety, and Tolerability of Two Fixed Dose Combinations of Aclidinium Bromide/Formoterol Fumarate, Aclidinium Bromide, Formoterol Fumarate and Placebo for 28- Weeks Treatment in Patients With Moderate to Severe, Stable Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy, Safety and Tolerability of Two Fixed Dose Combinations of Aclidinium Bromide/Formoterol Fumarate, Aclidinium Bromide, Formoterol Fumarate and Placebo for 28-Weeks Treatment in Patients With Moderate to Severe, Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAC-MD-36
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Aclidinium bromide/formoterol Fixed-Dose Combination (FDC) high dose
  Interventions: Drug: Aclidinium bromide/formoterol Fixed-Dose Combination (FDC)
- 2 (Experimental): Aclidinium bromide/formoterol Fixed-Dose Combination (FDC) low dose
  Interventions: Drug: Aclidinium bromide/formoterol Fixed-Dose Combination (FDC)
- 3 (Active Comparator): Aclidinium bromide 400 μg
  Interventions: Drug: Aclidinium bromide
- 4 (Active Comparator): Formoterol Fumarate 12 μg
  Interventions: Drug: Formoterol Fumarate
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide/formoterol Fixed-Dose Combination (FDC) — Inhaled Aclidinium bromide/formoterol Fixed-Dose Combination (FDC) high dose, twice per day
  Arms: 1
Drug: Aclidinium bromide/formoterol Fixed-Dose Combination (FDC) — Inhaled Aclidinium bromide/formoterol Fixed-Dose Combination (FDC) low dose, twice per day
  Arms: 2
Drug: Aclidinium bromide — Inhaled Aclidinium bromide 400 μg, twice per day
  Arms: 3
Drug: Formoterol Fumarate — Inhaled Formoterol Fumarate 12 μg, twice per day
  Arms: 4
Drug: Placebo — Inhaled dose-matched placebo, twice per day
  Arms: 5

SUMMARY:
The purpose of this Phase III study is to evaluate the long-term safety and tolerability of two fixed-dose combinations of inhaled aclidinium bromide/formoterol fumarate, aclidinium bromide, formoterol fumarate and placebo in patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD). Long-term efficacy, pharmacoeconomic and health-related quality of life assessments will also be evaluated. This extension study will include a 28 week treatment period, followed by a four week follow up visit. All patients will remain in the same treatment group as for the lead-in study and continue on one of the four treatment arms or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the treatment phase of the lead-in study, LAC-MD-31
* Written informed consent obtained from the patient before the initiation of any study specific procedures
* No medical contraindication as judged by the PI
* Compliance with LAC-MD-31 study procedures and IP dosing.

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (208):
- United States (179):
  - Forest Investigative Site 1827, Anniston, Alabama
  - Forest Investigative Site 1920, Athens, Alabama
  - Forest Investigative Site 1162, Birmingham, Alabama
  - Forest Investigative Site 1493, Birmingham, Alabama
  - Forest Investigative Site 1937, Birmingham, Alabama
  - Forest Investigative Site 1824, Gulf Shores, Alabama
  - Forest Investigative Site 2088, Jasper, Alabama
  - Forest Investigative Site 1918, Scottsboro, Alabama
  - Forest Investigative Site 0909, Glendale, Arizona
  - Forest Investigative Site 1379, Phoenix, Arizona
  - Forest Investigative Site 1822, Anaheim, California
  - Forest Investigative Site 1483, Buena Park, California
  - Forest Investigative Site 1156, Fresno, California
  - Forest Investigative Site 1871, Lincoln, California
  - Forest Investigative Site 1873, Los Angeles, California
  - Forest Investigative Site 2064, Riverside, California
  - Forest Investigative Site 1427, Sacramento, California
  - Forest Investigative Site 1866, Sacramento, California
  - Forest Investigative Site 1125, San Diego, California
  - Forest Investigative Site 2009, San Diego, California
  - Forest Investigative Site 1374, Torrance, California
  - Forest Investigative Site 1813, Tustin, California
  - Forest Investigative Site 1883, Vista, California
  - Forest Investigative Site 1380, Golden, Colorado
  - Forest Investigative Site 1137, Pueblo, Colorado
  - Forest Investigative Site 1327, Wheat Ridge, Colorado
  - Forest Investigative Site 1976, Waterbury, Connecticut
  - Forest Investigative Site 1821, Bay Pines, Florida
  - Forest Investigative Site 1154, Brandon, Florida
  - Forest Investigative Site 1944, Brandon, Florida
  - Forest Investigative Site 1364, Clearwater, Florida
  - Forest Investigative Site 1152, Clearwater, Florida
  - Forest Investigative Site 1875, Clearwater, Florida
  - Forest Investigative Site 1811, Covington, Florida
  - Forest Investigative Site 0670, DeLand, Florida
  - Forest Investigative Site 1516, Edgewater, Florida
  - Forest Investigative Site 0990, Fort Lauderdale, Florida
  - Forest Investigative Site 1513, Hialeah, Florida
  - Forest Investigative Site 1854, Hialeah, Florida
  - Forest Investigative Site 1882, Hollywood, Florida
  - Forest Investigative Site 1543, Jacksonville, Florida
  - Forest Investigative Site 1416, Kissimmee, Florida
  - Forest Investigative Site 1167, Melbourne, Florida
  - Forest Investigative Site 1432, Miami, Florida
  - Forest Investigative Site 1819, Naples, Florida
  - Forest Investigative Site 1808, North Miami, Florida
  - Forest Investigative Site 1950, Oldsmar, Florida
  - Forest Investigative Site 1145, Ormond Beach, Florida
  - Forest Investigative Site 1094, Panama City, Florida
  - Forest Investigative Site 1803, Pembroke Pines, Florida
  - Forest Investigative Site 0974, Pensacola, Florida
  - Forest Investigative Site 1817, Sarasota, Florida
  - Forest Investigative Site 1874, St. Petersburg, Florida
  - Forest Investigative Site 2082, Tamarac, Florida
  - Forest Investigative Site 2053, Tampa, Florida
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1185, Winter Park, Florida
  - Forest Investigative Site 1860, Winter Park, Florida
  - Forest Investigative Site 1900, Atlanta, Georgia
  - Forest Investigative Site 0987, Austell, Georgia
  - Forest Investigative Site 1828, Canton, Georgia
  - Forest Investigative Site 1830, Marietta, Georgia
  - Forest Investigative Site 2089, Woodstock, Georgia
  - Forest Investigative Site 0679, Coeur d'Alene, Idaho
  - Forest Investigative Site 1858, Eagle, Idaho
  - Forest Investigative Site 1095, Normal, Illinois
  - Forest Investigative Site 1912, Normal, Illinois
  - Forest Investigative Site 2051, River Forest, Illinois
  - Forest Investigative Site 2033, Bowling Green, Kentucky
  - Forest Investigative Site 2085, Fort Mitchell, Kentucky
  - Forest Investigative Site 0539, Lexington, Kentucky
  - Forest Investigative Site 1478, Louisville, Kentucky
  - Forest Investigative Site 1519, Owensboro, Kentucky
  - Forest Investigative Site 1430, New Orleans, Louisiana
  - Forest Investigative Site 1812, Opelousas, Louisiana
  - Forest Investigative Site 1814, Bangor, Maine
  - Forest Investigative Site 1924, Baltimore, Maryland
  - Forest Investigative Site 1872, Wheaton, Maryland
  - Forest Investigative Site 1570, Fall River, Massachusetts
  - Forest Investigative Site 1852, Fall River, Massachusetts
  - Forest Investigative Site 1431, No. Dartmouth, Massachusetts
  - Forest Investigative Site 1892, Ann Arbor, Michigan
  - Forest Investigative Site 1342, Stevensville, Michigan
  - Forest Investigative Site 1487, Troy, Michigan
  - Forest Investigative Site 1128, Edina, Minnesota
  - Forest Investigative Site 1527, Fridley, Minnesota
  - Forest Investigative Site 2041, Minneapolis, Minnesota
  - Forest Investigative Site 1124, Minneapolis, Minnesota
  - Forest Investigative Site 1619, Plymouth, Minnesota
  - Forest Investigative Site 1118, Rochester, Minnesota
  - Forest Investigative Site 1884, Olive Branch, Mississippi
  - Forest Investigative Site 1602, Kansas City, Missouri
  - Forest Investigative Site 1587, N. Chesterfield, Missouri
  - Forest Investigative Site 2079, Saint Charles, Missouri
  - Forest Investigative Site 1856, Springfield, Missouri
  - Forest Investigative Site 1867, Springfield, Missouri
  - Forest Investigative Site 1399, St Louis, Missouri
  - Forest Investigative Site 1599, St Louis, Missouri
  - Forest Investigative Site 1831, Bozeman, Montana
  - Forest Investigative Site 1400, Missoula, Montana
  - Forest Investigative Site 1609, Bellevue, Nebraska
  - Forest Investigative Site 1948, Fremont, Nebraska
  - Forest Investigative Site 1815, Lincoln, Nebraska
  - Forest Investigative Site 1363, Omaha, Nebraska
  - Forest Investigative Site 1907, Omaha, Nebraska
  - Forest Investigative Site 1911, Omaha, Nebraska
  - Forest Investigative Site 1908, Omaha, Nebraska
  - Forest Investigative Site 1804, Omaha, Nebraska
  - Forest Investigative Site 1807, Henderson, Nevada
  - Forest Investigative Site 1834, Las Vegas, Nevada
  - Forest Investigative Site 1562, Las Vegas, Nevada
  - Forest Investigative Site 1559, Cherry Hill, New Jersey
  - Forest Investigative Site 1923, Hackensack, New Jersey
  - Forest Investigative Site 1949, Albuquerque, New Mexico
  - Forest Investigative Site 1151, Great Neck, New York
  - Forest Investigative Site 1489, Larchmont, New York
  - Forest Investigative Site 550, New York, New York
  - Forest Investigative Site 1425, New York, New York
  - Forest Investigative Site 2098, Rochester, New York
  - Forest Investigative Site 1392, Charlotte, North Carolina
  - Forest Investigative Site 2035, Elizabeth City, North Carolina
  - Forest Investigative Site 1366, High Point, North Carolina
  - Forest Investigative Site 1153, Raleigh, North Carolina
  - Forest Investigative Site 1823, Salisbury, North Carolina
  - Forest Investigative Site 1891, Cadiz, Ohio
  - Forest Investigative Site 1134, Canton, Ohio
  - Forest Investigative Site 1885, Cincinnati, Ohio
  - Forest Investigative Site 1806, Cincinnati, Ohio
  - Forest Investigative Site 2028, Cincinnati, Ohio
  - Forest Investigative Site 1903, Cincinnati, Ohio
  - Forest Investigative Site 1361, Columbus, Ohio
  - Forest Investigative Site 1433, Columbus, Ohio
  - Forest Investigative Site 2090, Sylvania, Ohio
  - Forest Investigative Site 1530, Toledo, Ohio
  - Forest Investigative Site 1393, Zanesville, Ohio
  - Forest Investigative Site 1915, Oklahoma City, Oklahoma
  - Forest Investigative Site 1889, Bend, Oregon
  - Forest Investigative Site 2043, Medford, Oregon
  - Forest Investigative Site 1833, Altoona, Pennsylvania
  - Forest Investigative Site 1820, Downington, Pennsylvania
  - Forest Investigative Site 1423, Erie, Pennsylvania
  - Forest Investigative Site 1899, Langhorne, Pennsylvania
  - Forest Investigative Site 1443, Philadelphia, Pennsylvania
  - Forest Investigative Site 1863, Phoenixville, Pennsylvania
  - Forest Investigative Site 1146, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1449, Tipton, Pennsylvania
  - Forest Investigative Site 1862, Uniontown, Pennsylvania
  - Forest Investigative Site 1832, Cumberland, Rhode Island
  - Forest Investigative Site 1089, East Providence, Rhode Island
  - Forest Investigative Site 2072, Charleston, South Carolina
  - Forest Investigative Site 1905, Charleston, South Carolina
  - Forest Investigative Site 1802, Charleston, South Carolina
  - Forest Investigative Site 1914, Fort Mill, South Carolina
  - Forest Investigative Site 1913, Gaffney, South Carolina
  - Forest Investigative Site 1121, Spartanburg, South Carolina
  - Forest Investigative Site 1957, Brentwood, Tennessee
  - Forest Investigative Site 1526, Fayetteville, Tennessee
  - Forest Investigative Site 1440, Arlington, Texas
  - Forest Investigative Site 1879, Boerne, Texas
  - Forest Investigative Site 1861, Carrollton, Texas
  - Forest Investigative Site 1816, Corsicana, Texas
  - Forest Investigative Site 1890, Dallas, Texas
  - Forest Investigative Site 1332, El Paso, Texas
  - Forest Investigative Site 2012, Fort Worth, Texas
  - Forest Investigative Site 1951, Houston, Texas
  - Forest Investigative Site 1091, McKinney, Texas
  - Forest Investigative Site 1826, Plano, Texas
  - Forest Investigative Site 1895, San Antonio, Texas
  - Forest Investigative Site 1936, Salt Lake City, Utah
  - Forest Investigative Site 1330, South Burlington, Vermont
  - Forest Investigative Site 1945, Newport News, Virginia
  - Forest Investigative Site 1404, Norfolk, Virginia
  - Forest Investigative Site 1120, Bellingham, Washington
  - Forest Investigative Site 1977, Spokane, Washington
  - Forest Investigative Site 1878, Spokane, Washington
  - Forest Investigative Site 1573, Spokane, Washington
  - Forest Investigative Site 0988, Tacoma, Washington
  - Forest Investigative Site 1870, Tacoma, Washington
  - Forest Investigative Site 1555, Morgantown, West Virginia
- Australia (11):
  - Forest Investigative Site 1991, New Lambton, New South Wales
  - Forest Investigative Site 1987, Redcliffe, Queensland
  - Forest Investigative Site 1973, Woolloongabba, Queensland
  - Forest Investigative Site 2253, Adelaide, South Australia
  - Forest Investigative Site 1981, Bedford Park, South Australia
  - Forest Investigative Site 1990, Daw Park, South Australia
  - Forest Investigative Site 2251, Toorak Gardens, South Australia
  - Forest Investigative Site 2250, Clayton, Victoria
  - Forest Investigative Site 1972, Fitzroy, Victoria
  - Forest Investigative Site 1986, Geelong, Victoria
  - Forest Investigative Site 1985, Parkville, Victoria
- Canada (10):
  - Forest Investigative Site 1904, Langley, British Columbia
  - Forest Investigative Site 905, Vancouver, British Columbia
  - Forest Investigative Site 0976, Winnipeg, Manitoba
  - Forest Investigative Site 1877, Sarina, Ontario
  - Forest Investigative Site 1896, Sarnia, Ontario
  - Forest Investigative Site 1171, Toronto, Ontario
  - Forest Investigative Site 2203, Toronto, Ontario
  - Forest Investigative Site 1952, Montreal, Quebec
  - Forest Investigative Site 1859, Québec, Quebec
  - Forest Investigative Site 0943, Saskatoon, Saskatchewan
- New Zealand (8):
  - Forest Investigative Site 1027, Auckland
  - Forest Investigative Site 1970, Christchurch
  - Forest Investigative Site 1967, Dunedin
  - Forest Investigative Site 1964, Dunedin
  - Forest Investigative Site 1968, Hamilton
  - Forest Investigative Site 1965, Tauranga
  - Forest Investigative Site 1980, Tauranga
  - Forest Investigative Site 1025, Wellington

REFERENCES:
- [Derived] D'Urzo A, Rennard S, Kerwin E, Donohue JF, Lei A, Molins E, Leselbaum A. A randomised double-blind, placebo-controlled, long-term extension study of the efficacy, safety and tolerability of fixed-dose combinations of aclidinium/formoterol or monotherapy in the treatment of chronic obstructive pulmonary disease. Respir Med. 2017 Apr;125:39-48. doi: 10.1016/j.rmed.2017.02.008. Epub 2017 Feb 16. PMID 28340861
- See also: lac-md-36-synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4062&filename=lac-md-36-synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 169 study centers, 160 in the United States, and 9 in Canada. The first patient was screened in April 2012 and the last patient visit was in June 2013
Pre-assignment Details: This was a double-blind, placebo- and active-controlled, 28-week treatment, extension study of the lead-in study, Study LAC-MD-31
  Those patients who chose to continue the treatment in the extension study and met the eligibility for the extension study remained on the same treatment as they were randomized to in the lead-in study
Groups:
- Placebo: Placebo administered BID by inhalation
- Aclidinium/Formoterol 400/12 μg: Aclidinium bromide 400 μg + formoterol fumurate 12 μg fixed dose combination (FDC) administered BID by inhalation
- Aclidinium/Formoterol 400/6 μg: Aclidinium bromide 400 μg + formoterol fumurate 6 μg fixed dose combination (FDC) administered BID by inhalation
- Aclidinium 400 μg: Aclidinium bromide 400 μg administered BID by inhalation
- Formoterol 12 μg: Formoterol fumurate 12 μg administered BID by inhalation
Period: Lead-in Study
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Started | 337 | 338 | 338 | 340 | 339
Completed | 236 | 272 | 276 | 268 | 270
Not Completed | 101 | 66 | 62 | 72 | 69
Not completed — Lost to Follow-up | 5 | 9 | 4 | 2 | 4
Not completed — Withdrawal by Subject | 22 | 11 | 12 | 24 | 11
Not completed — Protocol Violation | 19 | 10 | 12 | 13 | 21
Not completed — Lack of Efficacy | 20 | 5 | 4 | 8 | 10
Not completed — Adverse Event | 21 | 21 | 22 | 16 | 14
Not completed — Site termination/COPD exacerbation/other | 14 | 10 | 8 | 9 | 9
Period: Extension Study
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Started | 146 | 184 | 205 | 194 | 192
Completed | 121 | 155 | 179 | 165 | 160
Not Completed | 25 | 29 | 26 | 29 | 32
Not completed — Lost to Follow-up | 6 | 2 | 0 | 3 | 3
Not completed — Withdrawal by Subject | 7 | 6 | 11 | 8 | 14
Not completed — Protocol Violation | 0 | 4 | 3 | 4 | 3
Not completed — Lack of Efficacy | 2 | 3 | 3 | 2 | 2
Not completed — Adverse Event | 7 | 6 | 5 | 6 | 4
Not completed — Site termination/COPD exacerbation/other | 3 | 8 | 4 | 6 | 6

BASELINE CHARACTERISTICS:
Population: The Extension Safety Population defined as all patients from the lead-in study (LAC-MD-31) who signed informed consent at Visit 1 of this extension study (last visit of the lead-in study) and who took at least 1 dose of double-blind investigational product in this extension study
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Total
Number analyzed (Participants) | 146 | 182 | 204 | 194 | 192 | 918
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.6) | 63.7 (9.1) | 63.6 (9.2) | 62.9 (8.3) | 62.8 (8.7) | 63.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 94 | 84 | 90 | 102 | 435
  Male | 81 | 88 | 120 | 104 | 90 | 483

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients to Experience Any Treatment-emergent Adverse Event
Description: For each safety parameter, the last assessment made before the first dose of investigational product in the lead-in study (LAC MD-31) was used as the baseline for all analyses of that safety parameter in this extension study
Time Frame: Baseline of lead-in study to follow-up call 14±3 days after last dose of investigational product (up to Week 52)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- Aclidinium/Formmoterol 400/12 μg: Aclidinium bromide 400 μg + formoterol fumurate 12 μg fixed dose combination (FDC) administered BID by inhalation
Arm/Group | Placebo | Aclidinium/Formmoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 146 | 182 | 204 | 194 | 192
Percentage of participants | 56.8 | 65.9 | 61.3 | 67.5 | 64.6

2. Secondary Outcome: Percentage of Patients to Experience Potentially Clinically Significant Post-baseline Clinical Laboratory Values for Hematology, Chemistry or Urinalysis
Description: Potentially clinically significant change:
  >1.15 × upper limit of normal (ULN) for absolute cell count of basophils, eosinophils or monocytes, blood alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, total bilirubin, blood urea nitrogen, total cholesterol, creatine kinase, creatinine, gamma glutamyl transferase, lactate dehydrogenase, triglycerides or uric acid <0.85 x lower limit of normal (LLN) or > 1.15 ULN for hematocrit ratio, haemoglobin, lymphocytes or neutrophils absolute cell count, platelet count (thrombocytes), red or white blood cell count, calcium, fasting glucose, phosphorus, total protein, or urinary pH <0.95 x LLN or >1.05 x ULN for chloride, potassium, sodium Urinary glucose ≥0.015, blood or ketones or protein ≥1 or specific gravity >1.1 × ULN
  The last assessment made before the first dose of investigational product in the lead-in study was used as the baseline for all safety analyses in the extension study
Time Frame: Baseline of lead-in study to end of treatment (up to Week 52)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aclidinium/Formmoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 146 | 182 | 204 | 194 | 192
Percentage of participants | 32.9 | 41.2 | 35.3 | 32.5 | 38.5

3. Secondary Outcome: Percentage of Patients to Experience a Potentially Significant Post-baseline 12-lead ECG Value
Time Frame: Baseline of lead-in study to end of treatment (up to Week 52)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aclidinium/Formmoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 146 | 182 | 204 | 194 | 192
Percentage of participants
  QT interval change from baseline >30 msec | 53.4 | 53.8 | 55.9 | 60.4 | 48.4
  QT interval >480 msec | 3.4 | 3.8 | 2.9 | 2.6 | 4.7
  QTcB change from baseline >30 msec | 36.3 | 37.0 | 39.7 | 35.6 | 38.4
  QTcB >480 msec | 7.5 | 8.3 | 9.8 | 5.7 | 8.4
  QTcF change from baseline >30 msec | 27.4 | 28.7 | 30.4 | 27.8 | 30.2
  QTcF >480 msec | 2.1 | 0.6 | 1.0 | 0.5 | 2.6
  QRS interval ≥100 msec & ≥25% increase | 6.2 | 6.6 | 3.9 | 2.6 | 4.7
  PR interval ≥200 msec & ≥25% increase | 2.8 | 2.2 | 1.0 | 3.1 | 1.6
  Heart rate ≥110 bpm & ≥15% increase from baseline | 0.7 | 2.7 | 1.0 | 1.0 | 2.1
  Heart rate ≤50 bpm & ≥15% decrease from baseline | 11.0 | 6.0 | 8.3 | 7.2 | 4.7

4. Other Pre Specified Outcome: Change From Baseline in 1-hour Morning Post-dose Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline of lead-in study to Week 52 of treatment
Population: The Combined intent to treat (ITT) Population defined as all patients randomized to a treatment group who took at least 1 dose of double-blind investigational product in the lead-in study (LAC-MD-31) and who had a baseline assessment and at least 1 post-baseline assessment of forced expiratory volume in 1 second (FEV1) in LAC-MD-31
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 331 | 335 | 333 | 337 | 332
Liters | -0.086 (0.017) | 0.198 (0.015) | 0.166 (0.015) | 0.112 (0.015) | 0.109 (0.015)

5. Other Pre Specified Outcome: Change From Baseline in Morning Predose (Trough) Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline of lead-in study to Week 52 of treatment
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 331 | 335 | 333 | 337 | 332
Liters | -0.101 (0.017) | 0.038 (0.015) | 0.005 (0.015) | 0.030 (0.015) | 0.004 (0.015)

6. Other Pre Specified Outcome: Transition Dyspnea Index (TDI) Focal Score at End of Study
Description: The TDI measures the change from baseline in severity of breathlessness in symptomatic patients. The TDI contains a rating for 3 categories (functional impairment, magnitude of task, magnitude of effort). TDI scale ranges from -3 (major deterioration) to +3 (major improvement) including a 0 score to indicate "no change". The 3 categories are added to obtain a focal score ranging from -9 (including 0) to +9.
Time Frame: Baseline of lead-in study to Week 52 of treatment
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 331 | 335 | 333 | 337 | 332
Scores on a scale | 0.731 (0.277) | 1.812 (0.251) | 1.742 (0.235) | 1.596 (0.241) | 1.324 (0.246)

7. Other Pre Specified Outcome: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Total Score
Description: St George's Respiratory Questionnaire (SGRQ) measures COPD-specific health outcomes and consists of 3 dimension scores (symptom, activity and impact). SGRQ total score is the sum of these scores and ranges from 0 (best health status) to 100 (worst health status).
Time Frame: Baseline of lead-in study to Week 52 of treatment
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 331 | 335 | 333 | 337 | 332
Scores on a scale | -1.862 (0.945) | -3.646 (0.861) | -5.527 (0.819) | -4.306 (0.847) | -4.059 (0.853)

8. Secondary Outcome: Percentage of Patients to Experience Potentially Clinically Significant Post-baseline Vital Signs (Pulse Rate, Systolic or Diastolic Blood Pressure or Weight)
Description: Potentially clinically significant change:
  Systolic BP ≥180 mmHg and increase ≥20 mmHg from baseline or ≤90 mmHg and decrease ≥20 mmHg from baseline Diastolic BP ≥105 mmHg and increase ≥15 mmHg from baseline or ≤50 mmHg and decrease ≥15 mmHg from baseline Pulse rate ≥110 bpm and increase ≥15% from baseline or ≤50 bpm and decrease ≥15% from baseline Weight increase or decrease ≥7% from baseline
  The last assessment made before the first dose of investigational product in the lead-in study was used as the baseline for all safety analyses in the extension study
Time Frame: Baseline of lead-in study to end of treatment (up to Week 52)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Aclidinium/Formmoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Number analyzed (Participants) | 146 | 182 | 204 | 194 | 192
Percentage of participants | 27.4 | 24.2 | 18.6 | 22.2 | 24.5

ADVERSE EVENTS:
Time Frame: Follow-up call 14±3 days after end of treatment (Week 28±5 days)
Description: The Extension Safety Population defined as all patients from the lead-in study (LAC-MD-31) who signed informed consent at Visit 1 of this extension study (last visit of the lead-in study) and who took at least 1 dose of double-blind investigational product in this extension study
Arm/Group | Placebo | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg
Serious Adverse Events (participants affected / at risk) | 10/146 | 14/182 | 14/204 | 15/194 | 14/192
Other Adverse Events (participants affected / at risk) | 37/146 | 59/182 | 64/204 | 67/194 | 62/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=146) | Aclidinium/Formoterol 400/12 μg (N=182) | Aclidinium/Formoterol 400/6 μg (N=204) | Aclidinium 400 μg (N=194) | Formoterol 12 μg (N=192)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 1 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=146) | Aclidinium/Formoterol 400/12 μg (N=182) | Aclidinium/Formoterol 400/6 μg (N=204) | Aclidinium 400 μg (N=194) | Formoterol 12 μg (N=192)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 6 | 12 | 5
Nasopharyngitis (Infections and infestations) | 7 | 14 | 14 | 18 | 13
Urinary tract infection (Infections and infestations) | 8 | 15 | 13 | 8 | 11
Upper respiratory tract infection (Infections and infestations) | 8 | 5 | 8 | 9 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 | 37 | 45 | 44 | 46

LIMITATIONS AND CAVEATS:
The objective of this extension study was to assess long-term safety and tolerability. Thus efficacy assessments were considered only supportive to the lead-in study (LAC-MD-31), and were not categorized as primary, secondary, or additional

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Principal Investigator (PI) will be subject to mutual agreement between the PI and the sponsor